CLINICAL TRIAL: NCT05333237
Title: Ultrasound Assessment of Gastric Emptying After a Standardized High Calorie Liquid Meal in Adults: a Prospective Observational Double-blind Study
Brief Title: Gastric Emptying of High Calorie Liquid Meals
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of Vienna (Other)
Responsible Party: Principal Investigator, Razvan Bologheanu, Principal Investigator, Medical University of Vienna
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Other
Other Study IDs: 1700_2021
Record Dates: First submitted 2022-03-28; First posted 2022-04-18 (Actual); Last update posted 2022-08-12 (Actual); Status verified 2022-08

CONDITIONS: Gastric Emptying
Keywords: Preoperative fasting; Liquid meal; Gastric ultrasound
MeSH Terms: interventions — Dietary Fiber; Glucose; Water

STUDY DESIGN:
Intervention Model Description: 3 interventions will be administered in fasted healthy volunteers in a random sequence on 3 different days.
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- Sequence 123 (Experimental): In this study arm the following sequence of interventions will be administered:
  upon first study session, intervention #1 will be administered (Dietary Supplement: ProvideXtra Drink).
  upon second study session, intervention #2 will be administered (Dietary Supplement: Fresubin Energy Drink).
  upon third study session, intervention #3 will be administered (Dietary Supplement: Generic Glucose Solution).
  Interventions: Dietary Supplement: Intervention #1: ProvideXtra Drink; Dietary Supplement: Intervention #2: Fresubin Energy Drink; Dietary Supplement: Intervention #3: Generic Glucose Solution
- Sequence 132 (Experimental): In this study arm the following sequence of interventions will be administered:
  upon first study session, intervention #1 will be administered (Dietary Supplement: ProvideXtra Drink).
  upon second study session, intervention #3 will be administered (Dietary Supplement: Generic Glucose Solution).
  upon third study session, intervention #2 will be administered (Dietary Supplement: Fresubin Energy Drink).
  Interventions: Dietary Supplement: Intervention #1: ProvideXtra Drink; Dietary Supplement: Intervention #2: Fresubin Energy Drink; Dietary Supplement: Intervention #3: Generic Glucose Solution
- Sequence 213 (Experimental): In this study arm the following sequence of interventions will be administered:
  upon first study session, intervention #2 will be administered (Dietary Supplement: Fresubin Energy Drink).
  upon second study session, intervention #1 will be administered (Dietary Supplement: ProvideXtra Drink).
  upon third study session, intervention #3 will be administered (Dietary Supplement: Generic Glucose Solution).
  Interventions: Dietary Supplement: Intervention #1: ProvideXtra Drink; Dietary Supplement: Intervention #2: Fresubin Energy Drink; Dietary Supplement: Intervention #3: Generic Glucose Solution
- Sequence 231 (Experimental): In this study arm the following sequence of interventions will be administered:
  upon first study session, intervention #2 will be administered (Dietary Supplement: Fresubin Energy Drink).
  upon second study session, intervention #3 will be administered (Dietary Supplement: Fresubin Energy Drink).
  upon third study session, intervention #1 will be administered (Dietary Supplement: ProvideXtra Drink).
  Interventions: Dietary Supplement: Intervention #1: ProvideXtra Drink; Dietary Supplement: Intervention #2: Fresubin Energy Drink; Dietary Supplement: Intervention #3: Generic Glucose Solution
- Sequence 312 (Experimental): In this study arm the following sequence of interventions will be administered:
  upon first study session, intervention #3 will be administered (Dietary Supplement: Generic Glucose Solution).
  upon second study session, intervention #1 will be administered (Dietary Supplement: ProvideXtra Drink).
  upon third study session, intervention #2 will be administered (Dietary Supplement: Fresubin Energy Drink).
  Interventions: Dietary Supplement: Intervention #1: ProvideXtra Drink; Dietary Supplement: Intervention #2: Fresubin Energy Drink; Dietary Supplement: Intervention #3: Generic Glucose Solution
- Sequence 321 (Experimental): In this study arm the following sequence of interventions will be administered:
  upon first study session, intervention #3 will be administered (Dietary Supplement: Generic Glucose Solution).
  upon second study session, intervention #2 will be administered (Dietary Supplement: Fresubin Energy Drink).
  upon third study session, intervention #1 will be administered (Dietary Supplement: ProvideXtra Drink).
  Interventions: Dietary Supplement: Intervention #1: ProvideXtra Drink; Dietary Supplement: Intervention #2: Fresubin Energy Drink; Dietary Supplement: Intervention #3: Generic Glucose Solution

INTERVENTIONS:
Dietary Supplement: Intervention #1: ProvideXtra Drink — Fasted subjects will be offered 200 ml of ProvideXtra and will be asked to ingest it at a comfortable rate. Subsequent gastric ultrasound examinations will be performed half-hourly (up to 6 hours) to determine the volume of the gastric contents. The intervention ends when the stomach appears to be empty again on ultrasound.
  Other Names: fat-free, high-calorie drink containing hydrolised vegetal protein
Dietary Supplement: Intervention #2: Fresubin Energy Drink — Fasted subjects will be offered 200 ml of Fresubin Energy Drink and will be asked to ingest it at a comfortable rate. Subsequent gastric ultrasound examinations will be performed half-hourly to determine the volume of the gastric contents. The intervention ends when the stomach appears to be empty again on ultrasound.
  Other Names: high-calorie drink without fiber
Dietary Supplement: Intervention #3: Generic Glucose Solution — Fasted subjects will be offered the glucose solution and will be asked to ingest it at a comfortable rate. Subsequent gastric ultrasound examinations will be performed half-hourly (up to 6 hours) to determine the volume of the gastric contents. The intervention ends when the stomach appears to be empty again on ultrasound.
  Other Names: Solution reconstituted form 75 g glucose and 300 ml water

SUMMARY:
Perioperative fasting is an essential patient safety measure to reduce the risk of pulmonary aspiration of gastric contents, a rare but potentially catastrophic complication of anesthetic and airway management. Anesthesiologists' concern about aspiration and the increasing awareness towards the negative impact of prolonged restriction of oral intake have shaped the current fasting guidelines. However, due to the perceived safety of prolonged fasting and practical considerations, adoption of the fasting guidelines is suboptimal.

Gastric ultrasound is a quick, non-invasive method to evaluate gastric contents and aspiration risk. Gastric ultrasound can accurately discriminate between solid particles and fluid content, and mathematical models can reliably predict the volume of the gastric contents from the gastric antral area (GAA).

This project aims to use gastric ultrasound to provide new data that can support management strategies in perioperative patients, that ensure both a low aspiration risk and an adequate nutritional support.

The investigators will test the hypothesis that commercially available liquid meals can be safely used preoperatively. A pilot crossover, study on healthy volunteers will be conducted to determine the gastric emptying time of high-calorie drinks, as compared to clear fluid.

ELIGIBILITY:
Inclusion Criteria:

* ASA 1 and 2

Exclusion Criteria:

* Allergy or intolerance to any of the study products or the ingredients
* Previous esophageal, gastric, or duodeno-pancreatic surgery
* Gastric banding or large hiatal hernia
* mmobility
* Contraindication to right lateral positioning
* Gastrointestinal diseases and disturbances
* Participation in another, possibly interfering study
* Diabetes mellitus
* Pregnancy

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2022-03-28 (Actual); Primary Completion 2022-05-18 (Actual); Study Completion 2022-06-01 (Actual)

PRIMARY OUTCOMES:
Gastric emptying time | Repeated ultrasound examinations will be performed every 30 minutes after the ingestion of the study product up to 6 hours after ingestion to determine whether the stomach has completely emptied.
  Time since ingestion of any of the study products until an empty stomach can be determined on ultrasound

SECONDARY OUTCOMES:
Gastric volume at prespecified intervals after ingestions | Ultrasound examinations will be repeated every 30 minutes after the ingestion of the study product up to 6 hours and the gastric antrum area and the gastric antrum cross-sectional area will be measured to estimate the volume of the gastric content.
  The volume of the gastric content determined using ultrasound

CONTACTS AND LOCATIONS:
Overall Officials: Andreas Duma, MSc, Principal Investigator — Medical University of Vienna
Locations (1):
- Medical University Vienna, Vienna, Austria

IPD SHARING:
Plan to Share IPD: Yes
IPD will be accessed by the PI upon request.
Supporting Information: CSR, Analytic Code
Time Frame: Data will be available from the PI 10 years after study completion.

REFERENCES:
- [Background] Smith I, Kranke P, Murat I, Smith A, O'Sullivan G, Soreide E, Spies C, in't Veld B; European Society of Anaesthesiology. Perioperative fasting in adults and children: guidelines from the European Society of Anaesthesiology. Eur J Anaesthesiol. 2011 Aug;28(8):556-69. doi: 10.1097/EJA.0b013e3283495ba1. PMID 21712716
- [Background] Tacken MCT, van Leest TAJ, van de Putte P, Keijzer C, Perlas A. Ultrasound assessment of gastric volumes of thick fluids: Validating a prediction model. Eur J Anaesthesiol. 2021 Dec 1;38(12):1223-1229. doi: 10.1097/EJA.0000000000001465. PMID 33606419
- [Background] Perlas A, Mitsakakis N, Liu L, Cino M, Haldipur N, Davis L, Cubillos J, Chan V. Validation of a mathematical model for ultrasound assessment of gastric volume by gastroscopic examination. Anesth Analg. 2013 Feb;116(2):357-63. doi: 10.1213/ANE.0b013e318274fc19. Epub 2013 Jan 9. PMID 23302981
- [Background] Perlas A, Arzola C, Van de Putte P. Point-of-care gastric ultrasound and aspiration risk assessment: a narrative review. Can J Anaesth. 2018 Apr;65(4):437-448. doi: 10.1007/s12630-017-1031-9. Epub 2017 Dec 11. PMID 29230709
- [Background] Van de Putte P, Perlas A. Ultrasound assessment of gastric content and volume. Br J Anaesth. 2014 Jul;113(1):12-22. doi: 10.1093/bja/aeu151. Epub 2014 Jun 3. PMID 24893784